CLINICAL TRIAL: NCT04517149
Title: An Open-label, Phase 1/2 Trial of Gene Therapy 4D-125 in Males With X-linked Retinitis Pigmentosa (XLRP) Caused by Mutations in the RPGR Gene
Brief Title: 4D-125 in Patients With X-Linked Retinitis Pigmentosa (XLRP)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: 4D Molecular Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 4D-125-C001
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: X-Linked Retinitis Pigmentosa
Keywords: XLRP; Gene therapy
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Intervention Model Description: In Phase 1, up to 2 dose exploration cohorts will be enrolled; each cohort will initially recruit up to 3 patients to receive a single uniocular IVT injection of 4D-125 in a standard 3+3 design. The cohort will be expanded in the event of a dose limiting toxicity (DLT). Any cohort may be expanded by an additional 3 subjects (to a maximum of 12 patients) to provide additional safety information and/or to confirm the selected dose for expansion. Once the dose level has been selected, the Phase 2 Dose Expansion Cohort will be opened to dose an additional 6-12 adult patients, and includes a pediatric sub-population of up to 6 patients. For adult participants only, the contralateral eye may also be dosed with 4D-125 as a single dose, IVT injection provided the subject is eligible and provides consent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 4D-125 Dose Exploration (Experimental): Dose 1 and Dose 2
  4D-125 will be administered at the assigned dose level as a single dose, IVT injection on Day 1. The contralateral eye may also be dosed with 4D-125 as a single dose, IVT injection provided the subject is eligible and provides consent.
  Interventions: Biological: 4D-125 IVT Injection
- 4D-125 Dose Expansion (Experimental): 4D-125 will be administered at the assigned dose level as a single dose, IVT injection on Day 1 in both adults and pediatric participants. For adult participants only, the contralateral eye may also be dosed with 4D-125 as a single dose, IVT injection provided the subject is eligible and provides consent.
  Interventions: Biological: 4D-125 IVT Injection
- Observational (Other): Natural History
  Interventions: Other: Observational

INTERVENTIONS:
Biological: 4D-125 IVT Injection — 4D-125 drug product developed for gene therapy, which comprises an AAV capsid variant (4D-R100) carrying a codon-optimized human Retinitis Pigmentosa GTPase Regulator transgene.
  Arms: 4D-125 Dose Expansion; 4D-125 Dose Exploration
Other: Observational — Natural History
  Arms: Observational

SUMMARY:
This is a Phase 1/2 multicenter study with two parallel parts: an observational natural history cohort and an open-label, prospective interventional trial in males with non-syndromic X-linked retinitis pigmentosa (XLRP) due to mutations in the gene encoding retinitis pigmentosa GTPase regulator (RPGR).

DETAILED DESCRIPTION:
This Phase 1/2 study will gather data in an observational phase Natural History Cohort to further characterize and evaluate natural disease progression in male patients with genetically-confirmed X-linked retinitis pigmentosa (XLRP) caused by mutations in the gene encoding retinitis pigmentosa GTPase regulator (RPGR). The study will also evaluate the safety and tolerability, as assessed by frequency and severity of ocular and systemic adverse events, as well as preliminary clinical efficacy of a single intravitreal (IVT) injection of 4D-125 at two dose levels in this patient population in one or both eyes (the contralateral eye dose provided the subject is eligible and provides consent).

4D-125 has been developed as a gene replacement therapy for XLRP. After receiving 4D-125, patients will be followed for 24 months with continued safety follow-up and 36 additional months of long-term follow-up. Secondary endpoints will assess preliminary efficacy measures over time after 4D-125 administration.

ELIGIBILITY:
Natural History Key Inclusion Criteria:

* Male, ≥ 6 years of age at the time of informed consent
* Hemizygous non-syndromic RPGR mutation confirmed by genetic testing

Interventional Key Inclusion Criteria:

* Male, ≥12 years of age
* Hemizygous non-syndromic RPGR mutation confirmed by genetic testing
* Phase 1 Dose Exploration: At least one eye amenable to IVT injection and BCVA ≤ 78 ETDRS letters (~20/32) and ≥ 34 ETDRS letters (~20/200)
* Phase 2 Dose Expansion: At least one eye amenable to IVT injection AND both eyes must have BCVA ≥ 34 ETDRS letters (~20/200)

Key Exclusion Criteria (all cohorts)

* Patient has previously received any AAV treatment
* Pre-existing eye conditions or surgical complications that would preclude participation in an interventional clinical trial or interfere with the interpretation of study endpoints

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of TEAEs and serious adverse events (SAEs), including clinically significant changes in safety parameters | 24 months to 60 Months

CONTACTS AND LOCATIONS:
Overall Officials: Schonmei Lee, MD, Study Director — 4D Molecular Therapeutics
Locations (8):
- United States (8):
  - University of Colorado, Aurora, Colorado
  - Vitreo Retinal Associates, Gainesville, Florida
  - University of Michigan Kellogg Eye Center, Ann Arbor, Michigan
  - Columbia University Medical Center/Edward Harkness Eye Institute, New York, New York
  - Duke University Eye Center/Dept. of Ophthalmology, Durham, North Carolina
  - Casey Eye Institute, Oregon Health and Science University, Portland, Oregon
  - Retina Foundation of the Southwest, Dallas, Texas
  - University of Utah John A. Moran Eye Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No